CLINICAL TRIAL: NCT00031226
Title: Biomarkers of Oxidative Stress in LOOK AHEAD - Ancillary to LOOK AHEAD
Status: Completed | Type: Observational
Sponsor: Arizona State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 993; R01HL070300 (NIH)
Record Dates: First submitted 2002-02-27; First posted 2002-02-28 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Heart Diseases; Myocardial Infarction; Obesity; Diabetes Mellitus, Non-insulin Dependent; Cardiovascular Diseases; Diabetes Mellitus
MeSH Terms: conditions — Heart Diseases; Myocardial Infarction; Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus

SUMMARY:
To determine how weight loss achieved by intensive lifestyle intervention including diet and exercise alters lipoprotein oxidation/oxidative stress and antioxidant status in overweight diabetic individuals.

DETAILED DESCRIPTION:
BACKGROUND:

Overweight and diabetes increase risk of cardiovascular disease but the mechanism(s) that account for this effect remain to be clarified. Oxidation of low-density lipoprotein (LDL) is thought to contribute to atherosclerosis. Diabetes may increase oxidative stress, and this may contribute to increased risk of cardiovascular disease in diabetics. Caloric restriction and the initiation of exercise may increase oxidative stress in the short term and may thus adversely affect cardiovascular disease. Over the long term, metabolic adaptation may reduce oxidative stress. Such adaptation, together with beneficial changes in lipoprotein concentration, composition, and character, may allow expression of beneficial effects of weight loss on cardiovascular endpoints. However, the influence of weight loss on measures of lipoprotein oxidation/oxidative stress and antioxidant status in overweight diabetics has never been investigated.

The study is ancillary to the Look AHEAD clinical trial which is sponsored primarily by the National Institute of Diabetes and Digestive and Kidney Diseases and secondarily by the National Heart, Lung, and Blood Institute, the National Institute of Nursing Research, the Office of Research on Women's Health, the National Center on Minority Health and Health Disparities, and the Centers for Disease Control and Prevention. The Look AHEAD study is a multicenter, randomized clinical trial to examine the long-term effects of a lifestyle intervention designed to achieve and maintain weight loss in overweight diabetics. The study is in response to an initiative on Ancillary Studies in Heart, Lung, and Blood Disease Trials released in June, 2000.

DESIGN NARRATIVE:

The primary aim of this project is to determine the influence of intensive lifestyle intervention on lipoprotein oxidation as assessed by autoantibodies to oxidized low-density lipoprotein. Other complementary indices of oxidative stress, and antioxidant status as assessed by circulating concentrations of lipophilic antioxidants, will be compared between lifestyle intervention and community care (control) arms of the Look AHEAD study. Such comparisons will be performed both early after intervention and later when metabolic adaptation is expected. By contrasting subgroups defined by differential compliance to diet or exercise, by gender, menopausal status, ethnicity, and age, secondary aims will consider whether changes in lipoprotein oxidation/oxidative stress and antioxidant status differ between such subgroups. Other aims will consider whether differences in lipoprotein oxidation/oxidative stress among the above subgroups can be accounted for by differences in lipoprotein concentration, composition, or character, carbohydrate metabolism, or antioxidant status. The results of this study will provide a potential mechanistic explanation for differences in cardiovascular endpoints between intervention and community care groups.

ELIGIBILITY:
An estimated 308 obese, diabetic subjects. There will be 184 women (60%) and 55% minorities.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Schwenke — Arizona State University